CLINICAL TRIAL: NCT05028686
Title: Predicting Readmissions Using Omics, Biostatistical Evaluate and Artificial Intelligence
Acronym: PROBE AI
Status: Recruiting | Type: Observational
Sponsor: Institute for Clinical Evaluative Sciences (Other)
Collaborators: Ted Rogers Centre for Heart Research (Unknown); Peter Munk Cardiac Centre (Unknown); Vector Institute for Artificial Intelligence (Unknown)
Responsible Party: Principal Investigator, Douglas Lee, Senior Scientist, Institute for Clinical Evaluative Sciences
Other Study IDs: 4
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples are stored in a biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized heart failure cohort: Patients hospitalized with heart failure
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational cohort

SUMMARY:
This study is a prospective registry that aims to predict readmissions in patients with heart failure, using -omics, machine learning, patient reported outcomes, clinical data and other high-dimensional data sources.

DETAILED DESCRIPTION:
There is substantial need to better predict outcomes across the spectrum of heart failure (HF) phenotypes in order to provide more efficient care with greater precision. Specifically, no validated methods have been adopted to predict outcomes reflecting transitions in health status across the continuum of HF and changes in cardiac function. A key transition is hospitalization - either readmission or de novo cardiovascular hospital admission. This is a major unmet health care need, to be able to better predict who will require hospital admission.

Novel contributions of biomarkers, -omics, remote patient monitoring, and artificial intelligence (AI). It is anticipated that prediction of readmission and many other outcomes will be further improved by measurement of circulating biomarkers and by incorporating methods from AI including machine learning and probabilistic generative models that can incorporate the lens of how physicians and patients think. Machine learning that incorporates many different types of data, including physician interpretation and a broad array of biomarker/-omics molecular information can lead to significant improvements in predictive accuracy. Novel multimarker strategies coupled with machine learning may enable the ability of physicians to predict a range of outcomes (e.g., transitions in HF health status and LVEF) and refine clinical prediction models. Furthermore, the investigators will collect patient data, including patient reported outcome measures (PROMs), and physiological data (e.g. heart rate, blood pressure, and daily weights data) and integrate these data points into predictive models. The investigators will use the PROMs obtainable using Medly as a predictor of hospitalization, and as an outcome. In this proposal, the investigators will take advantage of recent advances in both deep and high throughput proteomics technologies to perform high-resolution analyses. These novel factors can be integrated into new electronic algorithms to improve HF care in the population.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 18 years or older admitted to hospital or seen in the emergency department with heart failure defined clinically
* The diagnosis will be guided by the Framingham criteria for HF and/or BNP. A BNP >400 will be defined as definite heart failure and BNP 100-400 classified as possible heart failure.
* Provides informed consent

Exclusion Criteria:

* Patients who cannot communicate due to dementia or severe cognitive deficits
* non-Ontario residents
* nursing home residents
* those who are not discharged home but are discharged to a skilled nursing facility (long-term care or chronic institution)
* those who are unable to communicate who do not have a proxy (e.g. spouse or close family member) to facilitate communication with the patient.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular readmission | 30 day
  Non-elective readmission to hospital for a cardiovascular cause
Heart failure readmission | 30 day
  Non-elective readmission to hospital for heart failure

SECONDARY OUTCOMES:
Mortality | 30-day
  All-cause death
Cardiovascular death | 30-day
  Death from cardiovascular causes
All-cause readmission | 30-day
  Non-elective readmission to hospital for a any reason

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No